CLINICAL TRIAL: NCT00435513
Title: Association Study of a SRD5A2 SNP and Transsexualism.
Brief Title: A Common Polymorphism of the SRD5A2 Gene is Not Associated With Male-to-Female and Female-to-Male Transsexualism
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Clemens Tempfer, MD, Medical University of Vienna
Other Study IDs: 000001
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Transsexualism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transsexual group: Female-to-male and male-to-female transsexuals
- Controls: Healthy blood donors

SUMMARY:
Genetic variations, i.e. polymorphisms, may be associated with gender dysphoria, e.g. transsexualism. This study aims to identify such variations.

DETAILED DESCRIPTION:
Context: Early developmental exposure of the brain to sex steroids may play a role in the etiology of transsexualism.

Objective: To assess the association between transsexualism and allele and genotype frequencies of the steroid 5-alpha reductase (SRD5A2) Val89Leu polymorphism.

Design and Patients: We performed a case-control study of 100 male-to-female (MtF) transsexuals, 47 female-to-male (FtM) transsexuals, 755 male controls, and 915 female controls. DNA was extracted from buccal swabs and genotypes were determined by polymerase chain reaction.

Results: SRD5A2 Val89Leu allele frequencies (SRD5A2 V: 137/200 [69%] and SRD5A2 L: 63/200 [31%] vs. SRD5A2 V: 1065/1510 [71%] and SRD5A2 L: 445/1510 [29%], respectively; p=0.6; Odds Ratio [OR] 1.10; 95% Confidence Interval [CI] 0.76-1.58) and genotype distributions (SRD5A2 V/V+V/L: 92/100 [92%] and L/L 8/100 [8%] vs. SRD5A2 V/V+V/L: 683/755 [91%] and L/L 72/755 [9%], respectively, p=0.7; OR 0.82; 95% CI 0.24-2.84) were not significantly different between MtF transsexuals and male controls. SRD5A2 Val89Leu allele frequencies (SRD5A2 V: 70/94 [74%] and SRD5A2 L: 24/94 [26%] vs. SRD5A2 V: 1253/1830 [69%] and SRD5A2 L: 573/1830 [31%], respectively; p=0.3; OR 0.75; 95% CI 0.45-1.26) and genotype distributions (SRD5A2 V/V+V/L: 44/47 [93%] and L/L 3/47 [7%] vs. SRD5A2 V/V+V/L: 823/915 [90%] and L/L 92/915 [10%], respectively, p=0.6; OR 0.61; 95% CI 0.11-3.32) were also not significantly different between FtM transsexuals and female controls. Of note, there was no gender-specific genotype distribution among controls.

Conclusions: The SRD5A2 Val89Leu polymorphism is not associated with transsexualism and is no candidate gene of this condition.

ELIGIBILITY:
Inclusion Criteria:

* transsexual individuals as defined by DSM IV criteria

Exclusion Criteria:

* unwillingness to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female-to-male transsexuals and male-to-female transsexuals
Sampling Method: Probability Sample
Enrollment: 1770 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Principal Investigator — Univ. of Vienna
Locations (1):
- University of Vienna, Vienna, Austria, Vienna, Vienna, Austria